CLINICAL TRIAL: NCT02124252
Title: Evaluation of a Community-Driven Cervical Cancer Prevention Strategy in Western Kenya
Brief Title: Community-Driven Cervical Cancer Prevention in Western Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00077442
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-01

CONDITIONS: Human Papilloma Virus Infection; Carcinoma in Situ of Uterine Cervix
Keywords: cervical cancer screening; human papillomavirus testing; Kenya; implementation science
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Women will be offered HPV testing within the health facilities in the communities randomized to this arm. Women who test HPV positive will be referred to care at the sub-district and district hospitals (current standard of care).
- Standard Intervention (Active Comparator): Women will be offered HPV-based cervical cancer screening followed by standard linkage to care for women who test positive (to subdistrict or district hospitals).
  Interventions: Behavioral: Community-based testing with standard linkage to care
- Enhanced Intervention (Active Comparator): Women will be offered HPV-based cervical cancer screening followed by enhanced linkage to care using the strategies determined in partnership with the key stakeholders in the communities.
  Interventions: Behavioral: Community-based HPV testing with enhanced linkage to care

INTERVENTIONS:
Behavioral: Community-based testing with standard linkage to care — Women will be offered HPV-based cervical cancer screening followed by standard linkage to care for women who test positive (to subdistrict or district hospitals).
  Arms: Standard Intervention
Behavioral: Community-based HPV testing with enhanced linkage to care — Women will be offered HPV-based cervical cancer screening followed by enhanced linkage to care using the strategies determined in partnership with the key stakeholders in the communities.
  Arms: Enhanced Intervention

SUMMARY:
There are many challenges to implementation of cervical cancer prevention in resource-limited countries, despite evidence based screening and treatment strategies. The investigators hypothesize that self-collected HPV specimens offered in a community health campaign setting will

ELIGIBILITY:
Inclusion Criteria:

* Female, ages 25-65 Willing to sign informed consent Lives in community where randomization arm is

Exclusion Criteria:

* Prior hysterectomy

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7200 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Reach of cervical cancer screening using self-collected HPV specimens in community health campaigns compared to clinics | 2 years
  The investigators will compare the number of women who uptake HPV testing in the community health campaign arms compared to the number who uptake HPV testing in the clinic-based arms.

SECONDARY OUTCOMES:
Determine the Efficacy of the cervical cancer prevention program | 4 years
  The investigators will compare the number of women accessing treatment for positive HPV results with standard linkage to care compared to the enhanced linkage to treatment strategy.

OTHER OUTCOMES:
Determine the cost-effectiveness | 4-5 years
  The investigators will determine the cost-effectiveness of the three strategies in this study: clinic-based testing with standard referral to care, community-health campaign testing w/ standard referral to care & community based testing w/ enhanced linkage to care.

CONTACTS AND LOCATIONS:
Overall Officials: Megan J Huchko, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Olwanda EE, Kahn JG, Choi Y, Islam JY, Huchko M. Comparison of the costs of HPV testing through community health campaigns versus home-based testing in rural Western Kenya: a microcosting study. BMJ Open. 2020 Oct 27;10(10):e033979. doi: 10.1136/bmjopen-2019-033979. PMID 33109637
- [Derived] Huchko M, Adewumi K, Oketch S, Saduma I, Bukusi E. 'I'm here to save my life': a qualitative study of experiences navigating a cryotherapy referral system for human papillomavirus-positive women in western Kenya. BMJ Open. 2019 Jul 24;9(7):e028669. doi: 10.1136/bmjopen-2018-028669. PMID 31345973
- [Derived] Swanson M, Ibrahim S, Blat C, Oketch S, Olwanda E, Maloba M, Huchko MJ. Evaluating a community-based cervical cancer screening strategy in Western Kenya: a descriptive study. BMC Womens Health. 2018 Jul 3;18(1):116. doi: 10.1186/s12905-018-0586-0. PMID 29970063
- [Derived] Shen J, Olwanda E, Kahn JG, Huchko MJ. Cost of HPV screening at community health campaigns (CHCs) and health clinics in rural Kenya. BMC Health Serv Res. 2018 May 25;18(1):378. doi: 10.1186/s12913-018-3195-6. PMID 29801496
- [Derived] Huchko MJ, Kahn JG, Smith JS, Hiatt RA, Cohen CR, Bukusi E. Study protocol for a cluster-randomized trial to compare human papillomavirus based cervical cancer screening in community-health campaigns versus health facilities in western Kenya. BMC Cancer. 2017 Dec 6;17(1):826. doi: 10.1186/s12885-017-3818-z. PMID 29207966
- [Derived] Huchko MJ, Ibrahim S, Blat C, Cohen CR, Smith JS, Hiatt RA, Bukusi E. Cervical cancer screening through human papillomavirus testing in community health campaigns versus health facilities in rural western Kenya. Int J Gynaecol Obstet. 2018 Apr;141(1):63-69. doi: 10.1002/ijgo.12415. Epub 2018 Jan 3. PMID 29197067